CLINICAL TRIAL: NCT02412878
Title: A Randomized, Open-label, Phase 3 Study in Subjects With Relapsed and Refractory Multiple Myeloma Receiving Carfilzomib in Combination With Dexamethasone, Comparing Once-weekly Versus Twice-weekly Carfilzomib Dosing
Brief Title: Once-weekly Versus Twice-weekly Carfilzomib in Combination With Dexamethasone in Adults With Relapsed and Refractory Multiple Myeloma
Acronym: ARROW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFZ014; 2014-005325-12 (EudraCT Number); 20140355 (Other: Amgen Study ID)
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Results first posted 2018-12-13 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; WW Domain-Containing Oxidoreductase; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Once-weekly Carfilzomib 20/70 mg/m² + Dexamethasone (Experimental): Participants received carfilzomib administered by intravenous (IV) infusion on days 1, 8, and 15 of each 28-day cycle (20 mg/m² on day 1 of cycle 1 and 70 mg/m² thereafter).
  Participants also received 40 mg dexamethasone IV or orally on days 1, 8, 15 and 22 for the first 8 cycles; starting with cycle 9, dexamethasone was administered only on days 1, 8, and 15.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone
- Twice-weekly Carfilzomib 20/27 mg/m² + Dexamethasone (Experimental): Participants received carfilzomib administered by IV infusion on days 1, 2, 8, 9, 15, and 16 of each 28-day cycle (20 mg/m² on days 1 and 2 of cycle 1 and 27 mg/m² thereafter).
  Participants also received 40 mg dexamethasone IV or orally on days 1, 8, 15 and 22 for the first 8 cycles; starting with cycle 9, dexamethasone was administered only on days 1, 8, and 15.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib was administered as an IV infusion
  Other Names: PR-171; PR171; Kyprolis® (carfilzomib) for Injection
Drug: Dexamethasone — Commercially available dexamethasone was obtained by the investigational site.

SUMMARY:
The purpose of the study is to compare the progression-free survival (PFS) of once-weekly carfilzomib dosing in combination with dexamethasone to twice-weekly carfilzomib dosing in combination with dexamethasone in adults with relapsed and refractory multiple myeloma, previously treated with bortezomib and an immunomodulatory agent (IMiD).

ELIGIBILITY:
Key Inclusion Criteria:

1. Relapsed multiple myeloma
2. Refractory multiple myeloma defined as meeting 1 or more of the following:

   * Nonresponsive to most recent therapy (stable disease only or PD while on treatment), or
   * Disease progression within 60 days of discontinuation from most recent therapy
3. At least 2 but no more than 3 prior therapies for multiple myeloma
4. Prior exposure to an immunomodulatory agent (IMiD)
5. Prior exposure to a proteasome inhibitor (PI)
6. Documented response of at least partial response (PR) to 1 line of prior therapy
7. Measurable disease with at least 1 of the following assessed within the 21 days prior to randomization:

   * Serum M-protein ≥ 0.5 g/dL
   * Urine M-protein ≥ 200 mg/24 hours
   * In subjects without detectable serum or urine M-protein, serum free light chain (SFLC) > 100 mg/L (involved light chain) and an abnormal serum kappa lambda ratio
8. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1
9. Left ventricular ejection fraction (LVEF) ≥ 40% within the 21 days prior to randomization
10. Adequate organ and bone marrow function within the 21 days prior to randomization defined by:

    * Bilirubin < 1.5 times the upper limit of normal (ULN)
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 times the ULN
    * Absolute neutrophil count (ANC) ≥ 1000/mm³ (screening ANC should be independent of growth factor support for ≥ 1 week)
    * Hemoglobin ≥ 8.0 g/dL (Use of erythropoietic stimulating factors and red blood cell [RBC] transfusion per institutional guidelines is allowed, however the most recent RBC transfusion may not have been done within 7 days prior to obtaining screening hemoglobin.)
    * Platelet count ≥ 50,000/mm³ (≥ 30,000/mm³ if myeloma involvement in the bone marrow is > 50%. Subjects should not have received platelet transfusions for at least 1 week prior to obtaining the screening platelet count.)
    * Calculated or measured creatinine clearance (CrCl) of ≥ 30 mL/min

Key Exclusion Criteria:

1. Waldenström macroglobulinemia
2. Multiple myeloma of Immunoglobin M (IgM) subtype
3. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
4. Plasma cell leukemia (> 2.0 × 10⁹/L circulating plasma cells by standard differential)
5. Myelodysplastic syndrome
6. Second malignancy within the past 5 years except:

   * Adequately treated basal cell or squamous cell skin cancer
   * Carcinoma in situ of the cervix
   * Prostate cancer < Gleason score 6 with stable prostate-specific antigen (PSA) over 12 months
   * Ductal breast carcinoma in situ with full surgical resection (i.e., negative margins)
   * Treated medullary or papillary thyroid cancer
   * Similar condition with an expectation of > 95% five-year disease-free survival
7. History of or current amyloidosis
8. Cytotoxic chemotherapy within the 28 days prior to randomization
9. Immunotherapy within the 21 days prior to randomization
10. Glucocorticoid therapy within the 14 days prior to randomization that exceeds a cumulative dose of 160 mg of dexamethasone or 1000 mg prednisone
11. Radiation therapy:

    * Focal therapy within the 7 days prior to randomization
    * Extended field therapy within the 21 days prior to randomization
12. Prior treatment with either carfilzomib or oprozomib
13. Known history of allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib)
14. Contraindication to dexamethasone or any of the required concomitant drugs or supportive treatments, including hypersensitivity to antiviral drugs, or intolerance to hydration due to pre-existing pulmonary or cardiac impairment
15. Active congestive heart failure (New York Heart Association [NYHA] Class III or IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, acute diffuse infiltrative pulmonary disease, pericardial disease, or myocardial infarction within 6 months prior to enrollment
16. Active infection within the 14 days prior to randomization requiring systemic antibiotics
17. Pleural effusions requiring thoracentesis within the 14 days prior to randomization
18. Ascites requiring paracentesis within the 14 days prior to randomization
19. Ongoing graft-versus-host disease
20. Uncontrolled hypertension or uncontrolled diabetes despite medication
21. Significant neuropathy (≥ Grade 3) within the 14 days prior to randomization
22. Known cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2019-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (132):
- United States (12):
  - Research Site, Scottsdale, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Research Site, Bethesda, Maryland
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Research Site, Rockville, Maryland
  - Maryland Oncology Hematology, P.A, Rockville, Maryland
  - Research Site, Hackensack, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Research Site, New York, New York
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Tyler, Texas
  - Blood and Cancer Center of East Texas, Tyler, Texas
- Australia (4):
  - Research Site, Darlinghurst, New South Wales
  - Research Site, Tweed Heads, New South Wales
  - Research Site, Waratah, New South Wales
  - Research Site, Box Hill, Victoria
- Belgium (5):
  - Research Site, Antwerp
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
- Canada (9):
  - Research Site, Calgary, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Czechia (5):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Ostrava-Poruba
  - Research Site, Prague
- Denmark (4):
  - Research Site, Aalborg
  - Research Site, Copenhagen
  - Research Site, Odense C
  - Research Site, Vejle
- Finland (3):
  - Research Site, Helsinki
  - Research Site, Tampere
  - Research Site, Turku
- France (9):
  - Research Site, Bayonne
  - Research Site, Brest
  - Research Site, Dijon
  - Research Site, Nantes
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Rennes
  - Research Site, Tours
- Germany (5):
  - Research Site, Cologne
  - Research Site, Leipzig
  - Research Site, München
  - Research Site, Rostock
  - Research Site, Tübingen
- Greece (2):
  - Research Site, Athens
  - Research Site, Pátrai
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Gyula
  - Research Site, Kaposvár
- Italy (13):
  - Research Site, Ancona
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Cagliari
  - Research Site, Catania
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Napoli
  - Research Site, Pavia
  - Research Site, Piacenza
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Torino
- Japan (21):
  - Research Site, Toyohashi, Aichi-ken
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Ogaki-shi, Gifu
  - Research Site, Maebashi, Gunma
  - Research Site, Shibukawa-shi, Gunma
  - Research Site, Sapporo, Hokkaido
  - Research Site, Isehara-shi, Kanagawa
  - Research Site, Kyoto, Kyoto
  - Research Site, Sendai, Miyagi
  - Research Site, Okayama, Okayama-ken
  - Research Site, Suita-shi, Osaka
  - Research Site, Kawagoe-shi, Saitama
  - Research Site, Utsunomiya, Tochigi
  - Research Site, Chuo-ku, Tokyo
  - Research Site, Koto-ku, Tokyo
  - Research Site, Shibuya-ku, Tokyo
  - Research Site, Tachikawa-shi, Tokyo
  - Research Site, Fukuoka
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Tokushima
- New Zealand (2):
  - Research Site, Christchurch
  - Research Site, Otahuhu, Auckland
- Norway (2):
  - Research Site, Oslo
  - Research Site, Trondheim
- Poland (10):
  - Research Site, Brzozów
  - Research Site, Chorzów
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Romania (2):
  - Research Site, Brasov
  - Research Site, Bucharest
- Spain (9):
  - Research Site, Seville, Andalusia
  - Research Site, Zaragoza, Aragon
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Salamanca, Castille and León
  - Research Site, Badalona, Catalonia
  - Research Site, Barcelona, Catalonia
  - Research Site, Girona, Catalonia
  - Research Site, Pamplona, Navarre
  - Research Site, Madrid
- Sweden (5):
  - Research Site, Gothenburg
  - Research Site, Helsingborg
  - Research Site, Lund
  - Research Site, Stockholm
  - Research Site, Uddevalla
- United Kingdom (6):
  - Research Site, Bournemouth
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Nottingham
  - Research Site, Sheffield
  - Research Site, Wolverhampton

REFERENCES:
- [Background] Moreau P, Mateos MV, Berenson JR, Weisel K, Lazzaro A, Song K, Dimopoulos MA, Huang M, Zahlten-Kumeli A, Stewart AK. Once weekly versus twice weekly carfilzomib dosing in patients with relapsed and refractory multiple myeloma (A.R.R.O.W.): interim analysis results of a randomised, phase 3 study. Lancet Oncol. 2018 Jul;19(7):953-964. doi: 10.1016/S1470-2045(18)30354-1. Epub 2018 Jun 1. PMID 29866475
- [Background] Facon T, Niesvizky R, Mateos MV, Siegel D, Rosenbaum C, Bringhen S, Weisel K, Ho PJ, Ludwig H, Kumar S, Wang K, Obreja M, Yang Z, Klippel Z, Mezzi K, Goldrick A, Tekle C, Dimopoulos MA. Efficacy and safety of carfilzomib-based regimens in frail patients with relapsed and/or refractory multiple myeloma. Blood Adv. 2020 Nov 10;4(21):5449-5459. doi: 10.1182/bloodadvances.2020001965. PMID 33166401
- [Background] Dimopoulos MA, Niesvizky R, Weisel K, Siegel DS, Hajek R, Mateos MV, Cavo M, Huang M, Zahlten-Kumeli A, Moreau P. Once- versus twice-weekly carfilzomib in relapsed and refractory multiple myeloma by select patient characteristics: phase 3 A.R.R.O.W. study subgroup analysis. Blood Cancer J. 2020 Mar 9;10(3):35. doi: 10.1038/s41408-020-0300-y. PMID 32152297
- [Background] Moreau P, Stewart KA, Dimopoulos M, Siegel D, Facon T, Berenson J, Raje N, Berdeja JG, Orlowski RZ, Yang H, Ma H, Klippel Z, Zahlten-Kumeli A, Mezzi K, Iskander K, Mateos MV. Once-weekly (70 mg/m2 ) vs twice-weekly (56 mg/m2 ) dosing of carfilzomib in patients with relapsed or refractory multiple myeloma: A post hoc analysis of the ENDEAVOR, A.R.R.O.W., and CHAMPION-1 trials. Cancer Med. 2020 May;9(9):2989-2996. doi: 10.1002/cam4.2945. Epub 2020 Feb 28. PMID 32108443
- [Background] Moreau P, Kumar S, Boccia R, Iida S, Goldschmidt H, Cocks K, Trigg A, Zahlten-Kumeli A, Yucel E, Panjabi SS, Dimopoulos M. Convenience, satisfaction, health-related quality of life of once-weekly 70 mg/m2 vs. twice-weekly 27 mg/m2 carfilzomib (randomized A.R.R.O.W. study). Leukemia. 2019 Dec;33(12):2934-2946. doi: 10.1038/s41375-019-0480-2. Epub 2019 May 15. PMID 31092895
- [Background] Kumar SK, Majer I, Panjabi S, Medhekar R, Campioni M, Dimopoulos MA. Cost-effectiveness of once weekly carfilzomib 70 mg/m2 plus dexamethasone in patients with relapsed and refractory multiple myeloma in the United States. Expert Rev Hematol. 2020 Jun;13(6):687-696. doi: 10.1080/17474086.2020.1746639. Epub 2020 Apr 6. PMID 32249621
- [Derived] Dimopoulos MA, Moreau P, Iida S, Huang SY, Takezako N, Chng WJ, Zahlten-Kumeli A, Sersch MA, Li J, Huang M, Lee JH. Outcomes for Asian patients with multiple myeloma receiving once- or twice-weekly carfilzomib-based therapy: a subgroup analysis of the randomized phase 3 ENDEAVOR and A.R.R.O.W. Trials. Int J Hematol. 2019 Oct;110(4):466-473. doi: 10.1007/s12185-019-02704-z. Epub 2019 Aug 6. PMID 31388932
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from September 2015 to August 2016 at 118 sites in Australia, New Zealand, Japan, North America, and Europe.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive a regimen consisting of either once-weekly or twice weekly carfilzomib in combination with dexamethasone.
  Randomization was stratified by International Staging System (ISS) stage (stage 1 vs stages 2 or 3), refractory to bortezomib treatment (yes vs no), and age (< 65 vs ≥ 65 years).
Groups:
- Twice-weekly Carfilzomib 20/27 mg/m² + Dexamethasone: Participants received carfilzomib administered by intravenous (IV) infusion on days 1, 2, 8, 9, 15, and 16 of each 28-day cycle (20 mg/m² on days 1 and 2 of cycle 1 and 27 mg/m² thereafter).
  Participants also received 40 mg dexamethasone IV or orally on days 1, 8, 15 and 22 for the first 8 cycles; starting with cycle 9, dexamethasone was administered only on days 1, 8, and 15.
- Once-weekly Carfilzomib 20/70 mg/m² + Dexamethasone: Participants received carfilzomib administered by IV infusion on days 1, 8, and 15 of each 28-day cycle (20 mg/m² on day 1 of cycle 1 and 70 mg/m² thereafter).
  Participants also received 40 mg dexamethasone IV or orally on days 1, 8, 15 and 22 for the first 8 cycles; starting with cycle 9, dexamethasone was administered only on days 1, 8, and 15.
Period: Overall Study
Arm/Group | Twice-weekly Carfilzomib 20/27 mg/m² + Dexamethasone | Once-weekly Carfilzomib 20/70 mg/m² + Dexamethasone
Started | 238 | 240
Received Carfilzomib | 235 | 238
Completed (Defined as participants who discontinued due to death or study closure) | 217 | 227
Not Completed | 21 | 13
Not completed — Withdrawal by Subject | 19 | 10
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Population: The intention-to-treat population consisted of all randomly assigned participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Twice-weekly Carfilzomib 20/27 mg/m² + Dexamethasone | Once-weekly Carfilzomib 20/70 mg/m² + Dexamethasone | Total
Number analyzed (Participants) | 238 | 240 | 478
Age, Continuous [Median (Full Range); unit: years] | 66.0 [35 to 83] | 66.0 [39 to 85] | 66.0 [35 to 85]
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 104 | 104 | 208
  65 - 74 years | 102 | 90 | 192
  75 - 84 years | 32 | 45 | 77
  ≥ 85 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 108 | 218
  Male | 128 | 132 | 260
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 226 | 235 | 461
  Unknown or Not Reported | 7 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 15 | 30 | 45
  Black or African American | 2 | 3 | 5
  White | 202 | 200 | 402
  Other | 9 | 4 | 13
  Missing | 10 | 3 | 13
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care, unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  Participants
    0 (Fully active) | 118 | 118 | 236
    1 (Restrictive but ambulatory) | 120 | 121 | 241
    2 (Ambulatory but unable to work) | 0 | 1 | 1
Stratification Factor: International Staging System (ISS) stage [Count of Participants; unit: Participants] — The International Staging System (ISS) for myeloma was published by the International Myeloma Working Group:
  * Stage I: β2-microglobulin (β2M) < 3.5 mg/L, albumin >= 3.5 g/dL
  * Stage II: β2M < 3.5 mg/L and albumin < 3.5 g/dL; or β2M 3.5 mg/L - 5.5 mg/L irrespective of the serum albumin
  * Stage III: β2M ≥ 5.5 mg/L
  Participants
    Stage 1 | 100 | 100 | 200
    Stage 2 or 3 | 138 | 140 | 278
Stratification Factor: Refractory to Bortezomib Treatment [Count of Participants; unit: Participants] — Participants were classified as refractory to bortezomib in prior regimens if the data collected on prior multiple myeloma therapy indicated that any of the following criteria were met:
  1. Best Response to any regimen containing bortezomib was stable disease or progressive disease.
  2. Reason bortezomib was stopped was progression in any regimen.
  3. Date of relapse/progression was after start date and within 60 days after stop date of bortezomib in any regimen.
  Participants
    Yes | 88 | 88 | 176
    No | 150 | 152 | 302

OUTCOME MEASURES:

1. Secondary Outcome: Overall Response Rate
Description: Disease response was evaluated according to the IMWG-URC using a validated computer algorithm. Overall response rate was defined as the percentage of participants with a best overall response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR).
  sCR: As for CR, normal serum free light chain (SFLC) ratio and no clonal cells in bone marrow (BM).
  CR: No immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas and < 5% plasma cells in BM biopsy; VGPR: Serum and urine M-protein detectable by immunofixation but not electrophoresis or ≥ 90% reduction in serum M-protein with urine M-protein <100 mg/24 hours. A ≥ 50% reduction in the size of soft tissue plasmacytomas if present at baseline.
  PR: ≥ 50% reduction of serum M-protein and reduction in urine M-protein by ≥ 90% or to < 200 mg/24 hours. A ≥ 50% reduction in the size of soft tissue plasmacytomas if present at baseline.
Time Frame: Disease response was assessed every 28 days until progressive disease, up to the data cut-off date of 15 June 2017; median time on follow-up was 12.0 and 12.6 months in each treatment group respectively.
Population: Intent-to-treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Twice-weekly Carfilzomib 20/27 mg/m² + Dexamethasone | Once-weekly Carfilzomib 20/70 mg/m² + Dexamethasone
Number analyzed (Participants) | 238 | 240
percentage of participants | 40.8 [34.5 to 47.3] | 62.9 [56.5 to 69.0]
Statistical Analysis 1: Comparison: Twice-weekly Carfilzomib 20/27 mg/m² + Dexamethasone vs Once-weekly Carfilzomib 20/70 mg/m² + Dexamethasone; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Progression-free survival, overall response, and overall survival were tested using a fixed sequence hierarchical testing procedure to control the family-wise type I error rate below one-sided 0.025 level; One-sided p-value from CMH test stratified by the randomization factors (ISS stage at study entry, refractory to bortezomib treatment, and age); Odds Ratio (OR) = 2.485, 95% CI 2-sided [1.716 to 3.598] — Odds ratio (once weekly carfilzomib 20/70 mg/m²/ twice weekly carfilzomib 20/27 mg/m²) was calculated using the Mantel-Haenszel method stratified by the randomization stratification factors
Statistical Analysis 2: Comparison: Twice-weekly Carfilzomib 20/27 mg/m² + Dexamethasone vs Once-weekly Carfilzomib 20/70 mg/m² + Dexamethasone; Test type: Superiority; p < 0.0001, Fisher Exact; Odds Ratio (OR) = 2.466, 95% CI 2-sided [1.707 to 3.563] — Odds ratio (once weekly carfilzomib 20/70 mg/m²/ twice weekly carfilzomib 20/27 mg/m²) was calculated using the Mantel-Haenszel method

2. Primary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) was defined as the time from randomization to the earlier of disease progression or death due to any cause.
  Disease status was assessed at a central laboratory with serum and urine protein electrophoresis, immunofixation, serum-free light chain (SFLC) assay, bone marrow sample evaluation, serum calcium, plasmacytoma evaluation, and skeletal survey. Response and disease progression were determined using a validated computer algorithm based on the International Myeloma Working Group-Uniform Response Criteria (IMWG-URC).
  Median PFS was derived using the Kaplan-Meier method; participants still alive with no disease progression were censored at the time of their last disease assessment.
Time Frame: From randomization until the data cut-off date of 15 June 2017; median (minimum, maximum) follow-up time for PFS was 12.0 (0, 20) and 12.6 (0, 19) months in each treatment group respectively.
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Twice-weekly Carfilzomib 20/27 mg/m² + Dexamethasone | Once-weekly Carfilzomib 20/70 mg/m² + Dexamethasone
Number analyzed (Participants) | 238 | 240
months | 7.6 [5.8 to 9.2] | 11.2 [8.6 to 13.0]
Statistical Analysis 1: Comparison: Twice-weekly Carfilzomib 20/27 mg/m² + Dexamethasone vs Once-weekly Carfilzomib 20/70 mg/m² + Dexamethasone; To ensure proper control of type I error, analysis of PFS was performed under a group sequential design framework with the stopping boundaries constructed using the Lan-DeMets spending function with an O'Brien-Fleming approach. The inferential comparison between the 2 treatment groups for PFS used the 1-sided log-rank test stratified by the randomization stratification factors. A 1-sided p-value was compared against the prespecified adjusted alpha value of 0.011 to determine significance; Test type: Superiority; p = 0.0014, Log Rank — Progression-free survival, overall response rate, and overall survival were tested using a fixed sequence hierarchical testing procedure to control the family-wise type I error rate below one-sided 0.025 level; One-sided stratified log-rank test, stratified by the randomization factors (ISS stage at study entry, refractory to bortezomib treatment, and age); Hazard Ratio (HR) = 0.693, 95% CI 2-sided [0.544 to 0.883] — Hazard ratio (once weekly carfilzomib 20/70 mg/m²/ twice weekly carfilzomib 20/27 mg/m²) was estimated using a Cox proportional hazards model stratified by the randomization stratification factors
Statistical Analysis 2: Comparison: Twice-weekly Carfilzomib 20/27 mg/m² + Dexamethasone vs Once-weekly Carfilzomib 20/70 mg/m² + Dexamethasone; Test type: Superiority; p = 0.0033, Log Rank; One-sided unstratified log-rank test; Hazard Ratio (HR) = 0.720, 95% CI 2-sided [0.567 to 0.913] — Hazard ratio (once weekly carfilzomib 20/70 mg/m²/ twice weekly carfilzomib 20/27 mg/m²) was estimated using an unstratified Cox proportional hazards model

3. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) was defined as the time from randomization to death due to any cause.
  Median overall survival was derived using the Kaplan-Meier method; participants still alive were censored at the date last known to be alive.
Time Frame: From randomization until the data cut-off date of 15 June 2017; median (minimum, maximum) follow-up time for OS was 12.6 (0, 20) and 13.2 (0, 19) months in each treatment group respectively.
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Twice-weekly Carfilzomib 20/27 mg/m² + Dexamethasone | Once-weekly Carfilzomib 20/70 mg/m² + Dexamethasone
Number analyzed (Participants) | 238 | 240
months | NA [18.1 to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Twice-weekly Carfilzomib 20/27 mg/m² + Dexamethasone vs Once-weekly Carfilzomib 20/70 mg/m² + Dexamethasone; Test type: Superiority; p = 0.1070, Log Rank — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.800, 95% CI 2-sided [0.563 to 1.138] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Twice-weekly Carfilzomib 20/27 mg/m² + Dexamethasone vs Once-weekly Carfilzomib 20/70 mg/m² + Dexamethasone; Test type: Superiority; p = 0.1326, Log Rank; One-sided unstratified log-rank test; Hazard Ratio (HR) = 0.820, 95% CI 2-sided [0.578 to 1.164] — [estimate comment as in outcome 2, analysis 2]

4. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The severity of adverse events was graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03, where where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life-threatening; Grade 5 = Fatal.
  Treatment-related adverse events are adverse events considered related to at least 1 investigational product by the investigator, including those with unknown relationship.
Time Frame: From first dose of study drug up to 30 days after last dose, up to the end of study; median (minimum, maximum) duration of treatment was 29.1 (0.1, 156.3) weeks and 38.0 (0.1, 158.3) weeks in each treatment group respectively.
Population: All participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Twice-weekly Carfilzomib 20/27 mg/m² + Dexamethasone | Once-weekly Carfilzomib 20/70 mg/m² + Dexamethasone
Number analyzed (Participants) | 235 | 238
Participants
  Adverse events (AEs) | 230 | 233
  Adverse events Grade ≥ 3 | 152 | 181
  Serious adverse events | 102 | 118
  AEs leading to discontinuation of carfilzomib | 29 | 35
  AEs leading to discontinuation of dexamethasone | 31 | 40
  Fatal adverse events | 20 | 21
  Treatment-related adverse events (TRAEs) | 176 | 180
  Treatment-related adverse events Grade ≥ 3 | 82 | 108
  Serious treatment-related adverse events | 31 | 57
  TRAE leading to discontinuation of carfilzomib | 11 | 23
  TRAEs leading to discontinuation of dexamethasone | 13 | 29
  Fatal treatment-related adverse events | 3 | 5

5. Secondary Outcome: Plasma Carfilzomib Concentration During Cycle 2
Description: Concentrations of carfilzomib in plasma were measured using a validated assay method. The lower limit of quantification was 0.100 ng/mL.
Time Frame: Cycle 2 day 1 predose, 15 minutes after the start of infusion (once-weekly carfilzomib only), end of infusion, and 30 minutes after the end of infusion
Population: Participants at a subset of sites who participated in the sparse pharmacokinetic sampling, with available data at each time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Twice-weekly Carfilzomib 20/27 mg/m² + Dexamethasone | Once-weekly Carfilzomib 20/70 mg/m² + Dexamethasone
Number analyzed (Participants) | 36 | 55
ng/mL
  Predose | 36.2 (162) | 203 (1380)
  15 minutes after start of infusion: number analyzed (Participants) | 0 | 46
  15 minutes after start of infusion |  | 1370 (1410)
  End of infusion: number analyzed (Participants) | 10 | 51
  End of infusion | 1640 (1900) | 1130 (928)
  30 minutes after end of infusion: number analyzed (Participants) | 27 | 46
  30 minutes after end of infusion | 104 (293) | 480 (2300)

ADVERSE EVENTS:
Time Frame: All-cause mortality includes deaths that occurred from randomization until the end of study; median (minimum, maximum) follow-up time was 30.7 (0, 39) and 31.2 (0, 38) months in each treatment group respectively. Adverse events are reported from the first dose of study drug up to 30 days after last dose, as of the end of study; median (minimum, maximum) duration of treatment was 29.1 (0.1, 156.3) weeks and 38.0 (0.1, 158.3) weeks in each treatment group respectively.
Description: All-cause mortality is reported for all participants randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Twice-weekly Carfilzomib 20/27 mg/m² + Dexamethasone | Once-weekly Carfilzomib 20/70 mg/m² + Dexamethasone
All-Cause Mortality (participants affected / at risk) | 127/238 | 119/240
Serious Adverse Events (participants affected / at risk) | 102/235 | 118/238
Other Adverse Events (participants affected / at risk) | 204/235 | 217/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Twice-weekly Carfilzomib 20/27 mg/m² + Dexamethasone (N=235) | Once-weekly Carfilzomib 20/70 mg/m² + Dexamethasone (N=238)
Anaemia (Blood and lymphatic system disorders) | 8 | 4
Anaemia folate deficiency (Blood and lymphatic system disorders) | 1 | 0
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 1
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 3 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 3 | 3
Cardiac failure acute (Cardiac disorders) | 2 | 3
Cardiac failure congestive (Cardiac disorders) | 3 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 2 | 1
Retinal detachment (Eye disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Peritoneal haematoma (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 2
Catheter site vesicles (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Critical illness (General disorders) | 1 | 0
Death (General disorders) | 1 | 1
Disease progression (General disorders) | 3 | 2
Fatigue (General disorders) | 0 | 3
Papillitis (General disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 4
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 4 | 1
Bronchitis bacterial (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 4
Influenza (Infections and infestations) | 2 | 4
Lower respiratory tract infection (Infections and infestations) | 1 | 2
Lower respiratory tract infection viral (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 3
Lung infection pseudomonal (Infections and infestations) | 0 | 1
Neutropenic infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 1
Periodontitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 22 | 23
Pneumonia bacterial (Infections and infestations) | 3 | 3
Pneumonia haemophilus (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 3
Sepsis (Infections and infestations) | 3 | 6
Septic shock (Infections and infestations) | 2 | 5
Spinal cord infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
Wound infection bacterial (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 1
Liver function test abnormal (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 3
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 4
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Urethral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Intracranial mass (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Bradyphrenia (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 8 | 12
Renal failure (Renal and urinary disorders) | 3 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Homicide (Social circumstances) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 4 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1
Drug intolerance (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Perineal abscess (Infections and infestations) | 1 | 0
Post procedural sepsis (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1
General physical condition abnormal (Investigations) | 1 | 0
Monoclonal immunoglobulin present (Investigations) | 0 | 1
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Twice-weekly Carfilzomib 20/27 mg/m² + Dexamethasone (N=235) | Once-weekly Carfilzomib 20/70 mg/m² + Dexamethasone (N=238)
Anaemia (Blood and lymphatic system disorders) | 73 | 69
Neutropenia (Blood and lymphatic system disorders) | 23 | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 19 | 30
Constipation (Gastrointestinal disorders) | 22 | 21
Diarrhoea (Gastrointestinal disorders) | 51 | 53
Nausea (Gastrointestinal disorders) | 30 | 38
Vomiting (Gastrointestinal disorders) | 17 | 25
Asthenia (General disorders) | 29 | 29
Fatigue (General disorders) | 47 | 50
Oedema peripheral (General disorders) | 26 | 23
Pyrexia (General disorders) | 38 | 55
Bronchitis (Infections and infestations) | 25 | 31
Respiratory tract infection (Infections and infestations) | 23 | 18
Upper respiratory tract infection (Infections and infestations) | 28 | 39
Blood creatinine increased (Investigations) | 8 | 14
Neutrophil count decreased (Investigations) | 5 | 12
Platelet count decreased (Investigations) | 21 | 27
Decreased appetite (Metabolism and nutrition disorders) | 14 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 35
Bone pain (Musculoskeletal and connective tissue disorders) | 17 | 20
Muscle spasms (Musculoskeletal and connective tissue disorders) | 20 | 22
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 17
Headache (Nervous system disorders) | 25 | 28
Insomnia (Psychiatric disorders) | 49 | 39
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 44
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 27
Rash (Skin and subcutaneous tissue disorders) | 13 | 9
Hypertension (Vascular disorders) | 49 | 58
Cataract (Eye disorders) | 13 | 14
Chest pain (General disorders) | 4 | 12
Influenza (Infections and infestations) | 9 | 13
Nasopharyngitis (Infections and infestations) | 30 | 35
Pneumonia (Infections and infestations) | 5 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT02412878/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/78/NCT02412878/SAP_001.pdf